CLINICAL TRIAL: NCT01715805
Title: A Phase 3, Double-Blind, Placebo-Controlled Study of Cariprazine as Adjunctive Therapy in Major Depressive Disorder
Brief Title: Efficacy, Safety and Tolerability of Cariprazine as an Adjunctive Treatment to Antidepressant Therapy (ADT) in Patients With Major Depressive Disorder (MDD)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Forest Laboratories (Industry)
Collaborators: Gedeon Richter Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: RGH-MD-72
Record Dates: First submitted 2012-10-25; First posted 2012-10-29 (Estimated); Results first posted 2019-08-28 (Actual); Last update posted 2019-08-28 (Actual); Status verified 2019-08

CONDITIONS: Major Depressive Disorder
Keywords: MDD; Major Depressive Disorder
MeSH Terms: conditions — Depressive Disorder, Major | interventions — cariprazine

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- Placebo + ADT Lead-in (Other): Antidepressant therapy (ADT) as prescribed by the investigator plus single-blind placebo for 8 weeks.
  Interventions: Drug: Placebo; Drug: Antidepressant Therapy (ADT)
- Placebo + ADT (Double-Blind) (Placebo Comparator): Following the 8 week ADT plus single blind placebo lead-in period participants were randomized to dose-matched placebo, once per day, oral administration plus ADT for 8 weeks (up to Week 16).
  Interventions: Drug: Placebo; Drug: Antidepressant Therapy (ADT)
- Cariprazine + ADT (Double-Blind) (Experimental): Following the 8 week ADT plus single blind placebo lead-in period participants were randomized to cariprazine, 1.5 to 4.5 milligrams (mg) per day, oral administration plus ADT for 8 weeks (up to Week 16).
  Interventions: Drug: Cariprazine; Drug: Antidepressant Therapy (ADT)
- Placebo + ADT (Continued Treatment) (Other): Following the 8 week ADT plus single blind placebo lead-in period, participants who were ADT responders continued treatment with ADT plus placebo for an additional 8 weeks.
  Interventions: Drug: Placebo; Drug: Antidepressant Therapy (ADT)

INTERVENTIONS:
Drug: Cariprazine — Cariprazine capsules 1.5 to 4.5 mg/day
  Arms: Cariprazine + ADT (Double-Blind)
Drug: Placebo — Dose-matched placebo capsule once per day
  Arms: Placebo + ADT (Continued Treatment); Placebo + ADT (Double-Blind); Placebo + ADT Lead-in
Drug: Antidepressant Therapy (ADT) — ADT such as bupropion, citalopram, desvenlafaxine, duloxetine, escitalopram, fluoxetine, sertraline, venlafaxine, paroxetine or vilazodone as prescribed by the physician.

SUMMARY:
The objective of this study is to evaluate the efficacy, safety and tolerability of cariprazine as an adjunctive treatment to antidepressant therapy (ADT) in patients with MDD

ELIGIBILITY:
Inclusion Criteria:

* Patients who have provided consent prior to any specific procedure
* Meet the The Diagnostic and Statistical Manual of Mental Disorders, 4th edition, text revision (DSM-IV-TR) criteria for Major Depressive Disorder (MDD)
* Have a minimum score of 20 on 17-Item Hamilton Depression (HAMD-17) rating scale at Visits 1 and 2

Exclusion Criteria:

* Patients who do not meet DSM-IV-TR criteria for MDD

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1022 (Actual)
Dates: Start 2012-11-15 (Actual); Primary Completion 2016-06-24 (Actual); Study Completion 2016-06-24 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Willie Earley, MD, Study Director — Allergan
Locations (85):
- United States (83):
  - Forest Investigative Site 032, Tucson, Arizona
  - Forest Investigative Site 018, Little Rock, Arkansas
  - Forest Investigative Site 029, Little Rock, Arkansas
  - Forest Investigative Site 084, Cerritos, California
  - Forest Investigative Site 085, Culver City, California
  - Forest Investigative Site 082, Garden Grove, California
  - Forest Investigative Site 022, Newport Beach, California
  - Forest Investigative Site 004, Oceanside, California
  - Forest Investigative Site 090, Rancho Mirage, California
  - Forest Investigative Site 078, Redlands, California
  - Forest Investigative Site 080, Redlands, California
  - Forest Investigative Site 007, San Diego, California
  - Forest Investigative Site 054, San Diego, California
  - Forest Investigative Site 031, Temecula, California
  - Forest Investigative Site 048, Denver, Colorado
  - Forest Investigative Site 037, Coral Springs, Florida
  - Forest Investigative Site 053, Fort Myers, Florida
  - Forest Investigative Site 023, Hallandale, Florida
  - Forest Investigative Site 071, Hialeah, Florida
  - Forest Investigative Site 006, Leesburg, Florida
  - Forest Investigative Site 026, Miami, Florida
  - Forest Investigative Site 075, Miami, Florida
  - Forest Investigative Site 027, North Miami, Florida
  - Forest Investigative Site 074, North Miami, Florida
  - Forest Investigative Site 036, Oakland Park, Florida
  - Forest Investigative Site 051, Orlando, Florida
  - Forest Investigative Site 044, South Miami, Florida
  - Forest Investigative Site 008, Tampa, Florida
  - Forest Investigative Site 019, Winter Park, Florida
  - Forest Investigative Site 060, Atlanta, Georgia
  - Forest Investigative Site 024, Atlanta, Georgia
  - Forest Investigative Site 017, Marietta, Georgia
  - Forest Investigative Site 047, Smyrna, Georgia
  - Forest Investigative Site 070, Chicago, Illinois
  - Forest Investigative Site 013, Hoffman Estates, Illinois
  - Forest Investigative Site 063, Libertyville, Illinois
  - Forest Investigative Site 062, Maywood, Illinois
  - Forest Investigative Site 072, Naperville, Illinois
  - Forest Investigative Site 010, Oak Brook, Illinois
  - Forest Investigative Site 068, Skokie, Illinois
  - Forest Investigative Site 061, Indianapolis, Indiana
  - Forest Investigative Site 042, Lafayette, Indiana
  - Forest Investigative Site 065, Overland Park, Kansas
  - Forest Investigative Site 073, New Orleans, Louisiana
  - Forest Investigative Site 049, Gaithersburg, Maryland
  - Forest Investigative Site 077, Rockville, Maryland
  - Forest Investigative Site 012, Rockville, Maryland
  - Forest Investigative Site 046, Boston, Massachusetts
  - Forest Investigative Site 045, Natick, Massachusetts
  - Forest Investigative Site 086, Saint Charles, Missouri
  - Forest Investigative Site 014, Toms River, New Jersey
  - Forest Investigative Site 058, Albuquerque, New Mexico
  - Forest Investigative Site 028, Brooklyn, New York
  - Forest Investigative Site 016, New York, New York
  - Forest Investigative Site 083, New York, New York
  - Forest Investigative Site 025, Staten Island, New York
  - Forest Investigative Site 076, The Bronx, New York
  - Forest Investigative Site 050, Durham, North Carolina
  - Forest Investigative Site 067, Bismarck, North Dakota
  - Forest Investigative Site 088, Canton, Ohio
  - Forest Investigative Site 089, Cincinnati, Ohio
  - Forest Investigative Site 011, Cincinnati, Ohio
  - Forest Investigative Site 015, Cincinnati, Ohio
  - Forest Investigative Site 055, Columbus, Ohio
  - Forest Investigative Site 066, Mason, Ohio
  - Forest Investigative Site 064, Middleburg Heights, Ohio
  - Forest Investigative Site 035, Oklahoma City, Oklahoma
  - Forest Investigative Site 038, Oklahoma City, Oklahoma
  - Forest Investigative Site 039, Oklahoma City, Oklahoma
  - Forest Investigative Site 003, Portland, Oregon
  - Forest Investigative Site 052, Allentown, Pennsylvania
  - Forest Investigative Site 059, Lincoln, Rhode Island
  - Forest Investigative Site 001, Charleston, South Carolina
  - Forest Investigative Site 079, Austin, Texas
  - Forest Investigative Site 005, Houston, Texas
  - Forest Investigative Site 087, The Woodlands, Texas
  - Forest Investigative Site 069, Wichita Falls, Texas
  - Forest Investigative Site 030, Orem, Utah
  - Forest Investigative Site 041, Charlottesville, Virginia
  - Forest Investigative Site 081, Bellevue, Washington
  - Forest Investigative Site 043, Seattle, Washington
  - Forest Investigative Site 056, Milwaukee, Wisconsin
  - Forest Investigative Site 057, Waukesha, Wisconsin
- Puerto Rico (2):
  - Forest Investigative Site 033, San Juan
  - Forest Investigative Site 034, San Juan

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 1022 patients participated in an 8 week open label antidepression therapy (ADT) + single blind placebo lead-in period. 530 patients who did not respond were randomized to receive ADT or cariprazine + ADT in the double-blind period and non-responders continued ADT + Placebo.
Period: Placebo + ADT Lead-in Period
Arm/Group | Placebo + ADT Lead-in | Placebo + ADT (Double-Blind) | Cariprazine + ADT (Double-Blind) | Placebo + ADT (Continued Treatment)
Started | 1022 | 0 | 0 | 0
Completed | 807 | 0 | 0 | 0
Not Completed | 215 | 0 | 0 | 0
Not completed — Adverse Event | 41 | 0 | 0 | 0
Not completed — Insufficient therapeutic response | 6 | 0 | 0 | 0
Not completed — Protocol Violation | 74 | 0 | 0 | 0
Not completed — Withdrawal of Consent | 49 | 0 | 0 | 0
Not completed — Lost to Follow-up | 34 | 0 | 0 | 0
Not completed — Site Terminated by Sponsor | 1 | 0 | 0 | 0
Not completed — Other Reason Not Specified | 10 | 0 | 0 | 0
Period: Double-Blind or Continued Treatment
Arm/Group | Placebo + ADT Lead-in | Placebo + ADT (Double-Blind) | Cariprazine + ADT (Double-Blind) | Placebo + ADT (Continued Treatment)
Started | 0 | 261 | 269 | 270
Double-Blind Safety Population | 0 | 258 | 269 | 0
Completed | 0 | 222 | 213 | 222
Not Completed | 0 | 39 | 56 | 48
Not completed — Study or Site Terminated by Sponsor | 0 | 0 | 0 | 1
Not completed — Adverse Event | 0 | 3 | 23 | 2
Not completed — Protocol Violation | 0 | 14 | 12 | 19
Not completed — Withdrawal of consent | 0 | 11 | 11 | 13
Not completed — Lost to Follow-up | 0 | 7 | 10 | 10
Not completed — Other Reason Not Specified | 0 | 1 | 0 | 3
Not completed — Did not ingest Double-Blind Treatment | 0 | 3 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Pre-Randomization Safety Population included all patients in the screened population who took at least 1 dose of prospective open-label ADT plus single-blind placebo during the prospective ADT lead-in period of the study.
Arm/Group | Placebo + ADT Lead-in
Number analyzed (Participants) | 1022
Age, Continuous [Mean (Standard Deviation); unit: years] | 44.1 (12.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 673
  Male | 349
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race: White | 741
  Race: Black or African American | 250
  Race: Asian | 18
  Race: American Indian or Alaska Native | 8
  Race: Native Hawaiian or Other Pacific Islander | 3
  Race: Other | 2
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Ethnicity: Hispanic or Latino | 234
  Ethnicity: Not Hispanic or Latino | 788

OUTCOME MEASURES:

1. Primary Outcome: Montgomery-Asberg Depression Rating Scale (MADRS) at Baseline in the Double-Blind Period
Description: The MADRS is a clinician-rated scale to assess depressive symptomatology during the past week. Patients are rated on 10 items to assess feelings of sadness, lassitude, pessimism, inner tension, suicidality, reduced sleep or appetite, difficulty concentrating and lack of interest. Each item is scored on a 7-point scale. A score of 0 indicates the absence of symptoms, and a score of 6 indicates symptoms of maximum severity for a total possible score of 0 to 60.
Time Frame: Baseline (Week 8)
Population: Double-blind Intent-to-Treat (ITT) Population included all participants in the double-blind safety population who had a randomization baseline assessment and at least 1 postbaseline assessment of the MADRS total score during the double-blind treatment period.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Placebo + ADT (Double-Blind) | Cariprazine + ADT (Double-Blind)
Number analyzed (Participants) | 258 | 267
score on a scale | 25.2 (6.1) | 25.4 (5.5)

2. Primary Outcome: Change From Baseline in Montgomery-Asberg Depression Rating Scale (MADRS) in the Double-Blind Period
Description: The MADRS is a clinician-rated scale to assess depressive symptomatology during the past week. Participants are rated on 10 items to assess feelings of sadness, lassitude, pessimism, inner tension, suicidality, reduced sleep or appetite, difficulty concentrating and lack of interest. Each item is scored on a 7-point scale. A score of 0 indicates the absence of symptoms, and a score of 6 indicates symptoms of maximum severity for a total possible score of 0 to 60. A negative change from Baseline indicates improvement. Mixed-effects model for repeated measures (MMRM) with treatment group, study center, visit, and treatment group-by-visit interaction as fixed effects, and the baseline value and baseline by-visit interaction as the covariates was used for analyses.
Time Frame: Baseline (Week 8) to Week 16
Population: Double-blind ITT Population included all participants in the double-blind safety population who had a randomization baseline assessment and at least 1 postbaseline assessment of the MADRS total score during the double-blind treatment period.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Placebo + ADT (Double-Blind) | Cariprazine + ADT (Double-Blind)
Number analyzed (Participants) | 258 | 267
score on a scale | -7.5 (0.5) | -7.7 (0.5)
Statistical Analysis 1: Comparison: Placebo + ADT (Double-Blind) vs Cariprazine + ADT (Double-Blind); Test type: Superiority; p = 0.7948, Mixed Models Analysis — MMRM with treatment group, study center, visit, and treatment group-by-visit interaction as fixed effects, and the baseline value and baseline by-visit interaction as the covariates was used for analyses; Least Squares Mean Difference (LSMD) = -0.2, 95% CI 2-sided [-1.6 to 1.2] — Cariprazine + ADT - Placebo + ADT

3. Secondary Outcome: Change From Baseline in Sheehan Disability Scale (SDS) Score in the Double-Blind Period
Description: The Sheehan Disability Scale (SDS) is a 3-item patient-rated questionnaire used to evaluate impairments in the domains of work, social life/leisure, and family life/home responsibility. All items are rated on an 11-point continuum from 0 (no impairment) to 10 (most severe). The 3 individual scores are summed for a total possible score of 0 (unimpaired) to 30 (highly impaired). A negative change from Baseline indicates improvement. MMRM with treatment group, study center, visit, and treatment group-by-visit interaction as fixed effects, and the baseline value and baseline by-visit interaction as the covariates was used for analyses.
Time Frame: Baseline (Week 8) to Week 16
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Placebo + ADT (Double-Blind) | Cariprazine + ADT (Double-Blind)
Number analyzed (Participants) | 258 | 267
score on a scale | -3.1 (0.5) | -3.7 (0.5)
Statistical Analysis 1: Comparison: Placebo + ADT (Double-Blind) vs Cariprazine + ADT (Double-Blind); Test type: Superiority; p = 0.2784, Mixed Models Analysis — [p-value comment as in outcome 2, analysis 1]; LSMD = -0.7, 95% CI 2-sided [-1.9 to 0.5] — Cariprazine +ADT - Placebo + ADT

ADVERSE EVENTS:
Time Frame: First dose of study drug up to 30 days past last dose of study drug (Up to 12 Weeks for the ADT Lead-In arm) and up to an additional 12 weeks for the Double-Blind and Continued Treatment arms
Description: Other Adverse Events at a threshold of >=2% were analyzed separately for Lead-in, Double-Blind and Continued Treatment arms.
Arm/Group | Placebo + ADT Lead-in | Placebo + ADT (Double-Blind) | Cariprazine + ADT (Double-Blind) | Placebo + ADT (Continued Treatment)
All-Cause Mortality (participants affected / at risk) | 0/1022 | 0/258 | 0/269 | 0/270
Serious Adverse Events (participants affected / at risk) | 9/1022 | 3/258 | 1/269 | 1/270
Other Adverse Events (participants affected / at risk) | 261/1022 | 50/258 | 101/269 | 14/270
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo + ADT Lead-in (N=1022) | Placebo + ADT (Double-Blind) (N=258) | Cariprazine + ADT (Double-Blind) (N=269) | Placebo + ADT (Continued Treatment) (N=270)
Gastroenteritis (Infections and infestations) | 1 | 0 | 0 | 0
Pneumonia (Infections and infestations) | 1 | 0 | 0 | 0
Fall (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Lower limb fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Traumatic liver injury (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Cholecystitis (Hepatobiliary disorders) | 1 | 0 | 0 | 0
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Syncope (Nervous system disorders) | 1 | 0 | 0 | 0
Suicidal ideation (Psychiatric disorders) | 1 | 0 | 1 | 0
Abortion spontaneous (Pregnancy, puerperium and perinatal conditions) | 1 | 0 | 0 | 0
Migraine (Nervous system disorders) | 0 | 1 | 0 | 0
Seizure (Nervous system disorders) | 0 | 1 | 0 | 0
Pancreatitis acute (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Cholelithiasis (Hepatobiliary disorders) | 0 | 1 | 0 | 0
Depression (Psychiatric disorders) | 0 | 0 | 1 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Confusional state (Psychiatric disorders) | 0 | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo + ADT Lead-in (N=1022) | Placebo + ADT (Double-Blind) (N=258) | Cariprazine + ADT (Double-Blind) (N=269) | Placebo + ADT (Continued Treatment) (N=270)
Nausea (Gastrointestinal disorders) | 91 | 10 | 17 | 0
Diarrhoea (Gastrointestinal disorders) | 57 | 0 | 0 | 0
Nasopharyngitis (Infections and infestations) | 0 | 0 | 0 | 14
Headache (Nervous system disorders) | 91 | 15 | 22 | 0
Somnolence (Nervous system disorders) | 0 | 3 | 14 | 0
Insomnia (Psychiatric disorders) | 68 | 18 | 22 | 0
Akathisia (Nervous system disorders) | 0 | 8 | 46 | 0
Restlessness (Psychiatric disorders) | 0 | 5 | 23 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
A disclosure restriction on the PI is that the sponsor can review results communications prior to public release and can embargo communications regarding trial results for a period that is less than or equal to 90 days from the time submitted to the sponsor for review. The sponsor cannot require changes to the communication and cannot extend the embargo.